CLINICAL TRIAL: NCT02080364
Title: Randomized, Double-blind, Placebo Controlled, Multi-center Registration Trial to Evaluate the Efficacy and Safety of Azeliragon (TTP488) in Patients With Mild Alzheimer's Disease Receiving Acetylcholinesterase Inhibitors and/or Memantine
Brief Title: Evaluation of the Efficacy and Safety of Azeliragon (TTP488) in Patients With Mild Alzheimer's Disease
Acronym: STEADFAST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not due to safety but due to a lack of efficacy at the 5 mg azeliragon dose.
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTP488-301
Record Dates: First submitted 2014-02-25; First posted 2014-03-06 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; RAGE; ADAS-cog; CDR-sb
MeSH Terms: conditions — Alzheimer Disease | interventions — azeliragon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azeliragon 5mg (Experimental): Azeliragon (TTP488) 5mg orally once daily for 18 months
  Interventions: Drug: Azeliragon
- Placebo (Placebo Comparator): Placebo orally once daily for 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azeliragon — Azeliragon 5mg administered orally, once daily for 18 months
  Other Names: TTP488
  Arms: Azeliragon 5mg
Drug: Placebo — Placebo administered orally, once daily for 18 months
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of azeliragon in patients with mild Alzheimer's disease. Patients will receive either azeliragon or placebo with a patient's participation lasting approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer Disease (AD) with documented evidence of progression of disease
* Mini Mental State Examination (MMSE) score of 21-26, inclusive
* Clinical Dementia Rating global score of 0.5 or 1
* Rosen-Modified Hachinski Ischemia Score less than or equal to 4
* Brain magnetic resonance imaging (MRI) consistent with the diagnosis of probable AD
* Concurrent use of cholinesterase inhibitor or memantine with stable dose for at least 3 months prior to randomization
* Caregiver willing to participate and be able to attend clinic visits with patient
* Ability to ingest oral medications

Exclusion Criteria:

* Significant neurological or psychiatric disease other than Alzheimer's disease
* Participants with evidence or history of severe drug allergies (resulting in dyspnea or severe rash).
* Any contraindications to MRI (e.g., clinically significant claustrophobia, non-removable ferromagnetic implants). Patients with contraindications to MRI may undergo computed tomography (CT) on approval by sponsor.
* Any contraindications to the FDG-PET study (e.g. allergy to any component of the FDG dose) in the cohort undergoing a PET scan.
* Previous exposure to investigational or non-investigational therapies for Alzheimer's disease within 6 months of screening
* History of cancer within the last 5 years except adequately treated cervical carcinoma in-situ, cutaneous basal cell or squamous cell cancer, or non-progressive prostate cancer not requiring treatment
* Women of childbearing potential
* Uncontrolled blood pressure and/or blood pressure above 160/100
* Prescription medical food intended for dietary management of the metabolic processes associated with Alzheimer's disease.
* Diagnosis or history of cerebrovascular stroke, severe carotid stenosis, cerebral hemorrhage, intracranial tumor, subarachnoid hemorrhage.
* Patients with unstable, uncontrolled diabetes (HbA1c > 7.7%) and those requiring insulin.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron H Burstein, PharmD, Study Director — vTv Therapeutics
Locations (102):
- United States (70):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Bellflower, California
  - Costa Mesa, California
  - Fullerton, California
  - Glendale, California
  - Imperial, California
  - Irvine, California
  - Laguna Hills, California
  - Long Beach, California
  - Orange, California
  - Riverside, California
  - San Bernardino, California
  - San Francisco, California
  - Santa Ana, California
  - Atlantis, Florida
  - Brooksville, Florida
  - Delray Beach, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Sarasota, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Chicago, Illinois
  - Fairway, Kansas
  - Prairie Village, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Newton, Massachusetts
  - Plymouth, Massachusetts
  - Quincy, Massachusetts
  - Hattiesburg, Mississippi
  - Creve Coeur, Missouri
  - Princeton, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Lake Success, New York
  - New York, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Shaker Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Media, Pennsylvania
  - Norristown, Pennsylvania
  - Plains, Pennsylvania
  - East Providence, Rhode Island
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Cordova, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Murray, Utah
  - Kirkland, Washington
  - Richland, Washington
- Australia (6):
  - Southport, Queensland
  - Caulfield, Victoria
  - Geelong, Victoria
  - Heidelberg West, Victoria
  - Nedlands, Western Australia
  - West Perth, Western Australia
- Canada (8):
  - Calgary, Alberta
  - Medicine Hat, Alberta
  - Kentville, Nova Scotia
  - Chatham, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Gatineau, Quebec
  - Greenfield Park, Quebec
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Christchurch, Canterbury, New Zealand
- South Africa (3):
  - Cape Town
  - Johannesburg
  - Saint George
- United Kingdom (11):
  - Glasgow
  - London
  - Manchester
  - Northampton
  - Oxford
  - Penarth
  - Preston
  - Sheffield
  - Southhampton
  - Swindon
  - Warrington

REFERENCES:
- See also: Related Info — http://www.livingsteadfast.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The A-Study was conducted from April 2015 through April 2018 in the United States and Canada.
  The B-Study was conducted from September 2016 through June 2018 in the United States, Canada, United Kingdom, Ireland, South Africa, Australia and New Zealand.
Pre-assignment Details: A total of 1733 subjects underwent screening procedures for determination of eligibility for participation across the A- and B- Studies. 880 subjects were eligible and were randomized and assigned to treatment groups.
Groups:
- A-Study: Azeliragon; B-Study: Azeliragon: Azeliragon 5 mg once daily
- A-Study: Placebo: Placebo once daily
- B-Study: Placebo: Placebo capsule once daily
Period: Baseline Period
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Started | 197 | 208 | 247 | 228
Completed | 195 | 206 | 246 | 228
Not Completed | 2 | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0
Period: Treatment Period
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Started | 195 | 206 | 246 | 228
Completed | 148 | 157 | 9 | 4
Not Completed | 47 | 49 | 237 | 224
Not completed — Adverse Event | 10 | 15 | 11 | 14
Not completed — Lost to Follow-up | 2 | 3 | 5 | 0
Not completed — Protocol Violation | 5 | 3 | 5 | 1
Not completed — Withdrawal by Subject | 16 | 16 | 15 | 10
Not completed — Study Terminated by Sponsor | 0 | 0 | 180 | 183
Not completed — Other | 14 | 12 | 21 | 16

BASELINE CHARACTERISTICS:
Population: Demographics and Baseline Characteristics were analyzed using the Safety Analysis Set. The Safety Analysis set includes all randomized subjects who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo | Total
Number analyzed (Participants) | 195 | 206 | 246 | 228 | 875
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (9.13) | 74.9 (7.96) | 74.9 (8.55) | 74.4 (8.64) | 74.7 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 91 | 107 | 107 | 402
  Male | 98 | 115 | 139 | 121 | 473
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 23 | 8 | 15 | 73
  Not Hispanic or Latino | 168 | 183 | 238 | 213 | 802
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 5 | 2 | 6 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 0 | 3
  Black or African American | 8 | 9 | 8 | 5 | 30
  White | 179 | 194 | 231 | 220 | 824
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 0 | 0 | 6 | 3 | 9
  Canada | 25 | 25 | 16 | 18 | 84
  United States | 170 | 181 | 163 | 144 | 558
  Ireland | 0 | 0 | 9 | 7 | 16
  South Africa | 0 | 0 | 24 | 22 | 46
  United Kingdom | 0 | 0 | 20 | 27 | 47
  Australia | 0 | 0 | 8 | 7 | 15
Apo E4 status [Count of Participants; unit: Participants]
  Heterozygous | 83 | 79 | 115 | 105 | 382
  Homozygous | 15 | 27 | 31 | 18 | 91
  Non-carrier | 95 | 98 | 96 | 99 | 388
  Not reported | 2 | 2 | 4 | 6 | 14
Education Level [Count of Participants; unit: Participants]
  High School | 61 | 65 | 86 | 79 | 291
  Other (trainings, certifications) | 15 | 14 | 8 | 6 | 43
  Some college | 32 | 33 | 34 | 31 | 130
  Associates Degree | 17 | 14 | 14 | 21 | 66
  Bachelor's Degree | 44 | 39 | 64 | 55 | 202
  Master's Degree | 21 | 26 | 29 | 25 | 101
  Doctoral Degree | 5 | 15 | 11 | 11 | 42
Background AD Medication [Count of Participants; unit: Participants]
  Memantine | 12 | 16 | 19 | 22 | 69
  Acetylcholinesterase inhibitor | 117 | 124 | 156 | 145 | 542
  Both Memantine and Acetylcholinesterase inhibitor | 65 | 66 | 71 | 60 | 262
  Not recorded | 1 | 0 | 0 | 1 | 2
Years since AD diagnosis [Mean (Standard Deviation); unit: years] | 2.41 (2.389) | 2.32 (2.414) | 2.05 (1.932) | 1.86 (1.871) | 2.14 (2.153)
Baseline MMSE [Mean (Standard Deviation); unit: units on a scale] — The MMSE is a brief 30-point test that is used to assess cognition (Folstein, 1975). It is commonly used to screen for dementia. In the time span of about 10 minutes, it samples various functions, including arithmetic, memory and orientation. Scores range from 0-30 with lower scores indicating greater cognitive impairment. Population: Baseline MMSE was not reported / not valid for some subjects; therefore, the number analyzed is smaller than overall number.
  units on a scale
    number analyzed (Participants) | 189 | 202 | 244 | 225 | 860
    (all) | 23.42 (2.733) | 23.22 (2.522) | 23.29 (2.513) | 23.41 (2.701) | 23.33 (2.611)
Baseline ADAS-cog [Mean (Standard Deviation); unit: units on a scale] — The ADAS-cog is a structured scale (approximately 40 minutes to complete) that evaluates memory, orientation, attention, reasoning, language and constructional praxis (Rosen, 1984). The ADAS-cog scoring range for the version used in this study is from 0 to 70, with higher scores indicating greater cognitive impairment. Population: Baseline ADAScog was not reported / not valid for some subjects; therefore, the number analyzed is smaller than overall number.
  units on a scale
    number analyzed (Participants) | 188 | 202 | 243 | 225 | 858
    (all) | 15.42 (5.186) | 15.51 (5.427) | 16.94 (5.623) | 16.08 (5.295) | 16.05 (5.424)
Baseline CDR-Sum of Boxes [Mean (Standard Deviation); unit: units on a scale] — The CDR scale is used as a global measure of dementia and is completed by a clinician in the setting of detailed knowledge of the individual patient collected from interviews with the patient and caregiver (Berg, 1988). The CDR describes 5 degrees of impairment in performance on each of 6 categories including memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Sum of box scores range from 0 to 18 with higher scores indicating greater cognitive impairment. Population: Baseline CDR-sb was not reported / not valid for some subjects; therefore, the number analyzed is smaller than overall number.
  units on a scale
    number analyzed (Participants) | 189 | 202 | 244 | 225 | 860
    (all) | 4.06 (1.747) | 4.07 (1.623) | 4.64 (1.585) | 4.5 (1.570) | 4.34 (1.645)
Baseline ADCS-ADL [Mean (Standard Deviation); unit: units on a scale] — The ADCS-ADL is an activity of daily living inventory developed by the ADCS to assess functional performance in participants with AD (Galasko et al., 1997). Informants are queried via a structured interview format as to whether participants attempted each item in the inventory during the preceding 4 weeks, as well as their level of performance. Scores range from 0-78 with lower scores indicating greater functional impairment. Population: Baseline ADCS-ADL was not reported / not valid for some subjects; therefore, the number analyzed is smaller than overall number.
  units on a scale
    number analyzed (Participants) | 189 | 202 | 244 | 225 | 860
    (all) | 67.62 (7.67) | 67.37 (8.56) | 66.25 (8.142) | 67.25 (7.568) | 67.08 (8.001)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog) Total Score
Description: The ADAS-cog is a structured scale (approximately 40 minutes to complete) that evaluates memory, orientation, attention, reasoning, language and constructional praxis (Rosen, 1984). The ADAS-cog scoring range for the version used in this study is from 0 to 70, with higher scores indicating greater cognitive impairment.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: Full Analysis Set (all randomized subjects who receive study medication and have at least one post-baseline efficacy assessment) with Month 18 (A-Study) or Month 12 (B-Study) data. B-Study excludes data from visits occurring after A-Study results announcement on 09 Apr 2018. ADAS-cog was not reported / not valid for some subject visits; therefore, the number analyzed is smaller than overall number.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 138 | 151 | 118 | 121
score on a scale | 3.8 (0.51) | 3.1 (0.49) | 3.4 (0.46) | 2.5 (0.46)
Statistical Analysis 1: Comparison: A-Study: Azeliragon vs A-Study: Placebo; Test type: Superiority; p = 0.3386, Mixed Models Analysis — p-value for comparison to Placebo
Statistical Analysis 2: Comparison: B-Study: Azeliragon vs B-Study: Placebo; Test type: Superiority; p = 0.1992, Mixed Models Analysis — p-value for compairons to Placebo

2. Primary Outcome: Change From Baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-sb)
Description: The CDR scale is used as a global measure of dementia and is completed by a clinician in the setting of detailed knowledge of the individual patient collected from interviews with the patient and caregiver (Berg, 1988). The CDR describes 5 degrees of impairment in performance on each of 6 categories including memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. CDR ratings are 0 for healthy individuals, 0.5 for questionable dementia and 1, 2 and 3 for mild, moderate and severe dementia as defined in the CDR scale. The scores for each category can also be summed and this is known as the sum of box score (CSR-SB). Sum of box scores range from 0 to 18 with higher scores indicating greater cognitive impairment.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: Full Analysis Set (all randomized subjects who receive study medication and have at least one post-baseline efficacy assessment) with Month 18 (A-Study) or Month 12 (B-Study) data. B-Study excludes data from visits occurring after A-Study results announcement on 09 Apr 2018. CDR-sb was not reported / not valid for some subject visits; therefore, the number analyzed is smaller than overall number.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 140 | 150 | 117 | 120
score on a scale | 1.4 (2.23) | 1.4 (1.85) | 1.3 (1.87) | 0.7 (1.4)
Statistical Analysis 1: Comparison: A-Study: Azeliragon vs A-Study: Placebo; Test type: Superiority; p = 0.9394, Mixed Models Analysis — p-value for comparison to Placebo
Statistical Analysis 2: Comparison: B-Study: Azeliragon vs B-Study: Placebo; Test type: Superiority; MMRM model does not converge. LS Mean and p-value are NA

3. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) Brain Volumetric Measures
Description: Percent of Total Hippocampus Atrophy to Intracranial Volume
Time Frame: Baseline and 18 months
Population: Number of subjects with paired Baseline and Month 18 MRIs
Measure: Least Squares Mean (Standard Error); unit: percentage of Total Hippocampus Atrophy
Arm/Group | Azeliragon 5mg | Placebo
Number analyzed (Participants) | 112 | 116
percentage of Total Hippocampus Atrophy | -0.016 (0.001) | -0.014 (0.001)

4. Secondary Outcome: Change From Baseline in the Normalized Mean Composite SUVR of the 5 Regions
Description: Extent and severity of brain hypometabolism was assessed centrally at Baseline and Month 18. SUVR PET was designed to make use of FreeSurfer-based segmentations of the brain obtained using the 3DT1 MRI. Following the methods published by Landau and Jagust (Landau SM, Annals of Neurology 2012) and described on the ADNI website (http://adni.loni.usc.edu/methods/pet-analysis-method/), regions were defined in native patient space on the 3DT1 MRI acquired at the Baseline visit and at Month 18 visit. An SUVR measure was computed regionally over five sub-regions (anterior/posterior cingulate, temporal, parietal, frontal and hippocampal areas), normalized to activity in the cerebral white matter. These sub-regions were selected to optimize sensitivity in longitudinal studies. This outcome measure presents the change from baseline in the normalized mean composite SUVR of the 5 regions. A negative change from baseline indicates a decrease (worsening) in brain glucose metabolism/utilization.
Time Frame: Baseline to 18 months
Population: Analyzed as part of an optional FDG-PET substudy
Measure: Least Squares Mean (Standard Error); unit: SUVR ratio
Arm/Group | Azeliragon 5mg | Placebo
Number analyzed (Participants) | 38 | 36
SUVR ratio | -0.0304 (0.0039) | -0.0342 (0.0039)

5. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study- Activities of Daily Living Inventory (ADCS-ADL)
Description: The ADCS-ADL is an activity of daily living inventory developed by the ADCS to assess functional performance in participants with AD (Galasko et al., 1997). Informants are queried via a structured interview format as to whether participants attempted each item in the inventory during the preceding 4 weeks, as well as their level of performance. Scores range from 0-78 with lower scores indicating greater functional impairment.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: Full Analysis Set (all randomized subjects who receive study medication and have at least one post-baseline efficacy assessment) with Month 18 (A-Study) or Month 12 (B-Study) data. B-Study excludes data from visits occurring after A-Study results announcement on 09 Apr 2018. ADCS-ADL was not reported / not valid for some subject visits; therefore, the number analyzed is smaller than overall number.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 141 | 152 | 121 | 122
score on a scale | -5.1 (8.63) | -3.2 (8.92) | -5.4 (8.85) | -2.8 (7.83)

6. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE)
Description: The MMSE is a brief 30-point test that is used to assess cognition (Folstein, 1975). It is commonly used to screen for dementia. In the time span of about 10 minutes, it samples various functions, including arithmetic, memory and orientation. Scores range from 0-30 with lower scores indicating greater cognitive impairment.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: Full Analysis Set (all randomized subjects who receive study medication and have at least one post-baseline efficacy assessment) with Month 18 (A-Study) or Month 12 (B-Study) data. B-Study excludes data from visits occurring after A-Study results announcement on 09 Apr 2018. MMSE was not reported / not valid for some subject visits; therefore, the number analyzed is smaller than overall number.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 142 | 153 | 121 | 121
score on a scale | -2.1 (3.55) | -2.0 (3.25) | -2.1 (3.25) | -1.8 (3.29)

7. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI)
Description: The NPI is a well-validated, reliable, multi-item instrument to assess psychopathology in AD based on an interview with the caregiver (Cummings et al, 1994). It evaluates both the frequency and severity of 12 behavioral areas including delusions, hallucinations, dysphoria (depression) anxiety, agitation/aggression, euphoria, disinhibition, irritability, lability, apathy, aberrant motor behavior, appetite and eating changes and night-time behaviors.
  Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously) as well as severity (1= mild, 2 = moderate, 3 = severe). Distress is rated by the study partner or caregiver and ranges from 0 (no distress) to 5 (very severe or extreme). The overall score and the score for each subscale are the product of severity and frequency. Scores range from 0-144 with higher scores indicating a greater presence of neuropsychiatric symptoms.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: Full Analysis Set (all randomized subjects who receive study medication and have at least one post-baseline efficacy assessment) with Month 18 (A-Study) or Month 12 (B-Study) data. B-Study excludes data from visits occurring after A-Study results announcement on 09 Apr 2018. NPI was not reported / not valid for some subject visits; therefore, the number analyzed is smaller than overall number.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 142 | 152 | 121 | 122
score on a scale | -0.2 (9.77) | 1.3 (11.53) | 2.3 (11.24) | 0.0 (10.67)

8. Secondary Outcome: Change From Baseline in Dementia Quality of Life (DEMQOL)
Description: The DEMQOL-Proxy questionnaire is a validated and reliable questionnaire that is interview administered and completed by the caregiver about the patient's health related quality of life (Smith et al, 2005). It consists of 31 items representing 5 domains (daily activities and looking after yourself, health and well-being, cognitive functioning, social relationships, and self-concept) and takes approximately 20 minutes to complete. Scores range 31-124 with higher scores indicate better health related quality of life.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: Full Analysis Set (all randomized subjects who receive study medication and have at least one post-baseline efficacy assessment) with Month 18 (A-Study) or Month 12 (B-Study) data. DEMQOL was not reported / not valid for some subject visits; therefore, the number analyzed is smaller than overall number.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 142 | 152 | 179 | 187
score on a scale | 0.0 (10.2) | -1.2 (9.38) | -0.1 (10.55) | -0.8 (11.70)

9. Secondary Outcome: Change From Baseline in Continuous Oral Word Association Task (COWAT)
Description: The COWAT is a measure of verbal fluency in which the participant is asked to generate orally as many words as possible that begin with the letters "F", "A", and "S", excluding proper names and different forms of the same word. (Borkowski, 1967, Loonstra 2001) For each letter, the participant is allowed one minute to generate the words. Performance is measured by the total number of correct words produced summed across the three letters. Perseverations (i.e., repetitions of a correct word) and intrusions (i.e., words not beginning with the designated letter) are noted.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: Full Analysis Set (all randomized subjects who receive study medication and have at least one post-baseline efficacy assessment) with Month 18 (A-Study) or Month 12 (B-Study) data. NPI was not reported / not valid for some subject visits; therefore, the number analyzed is smaller than overall number.
Measure: Mean (Standard Deviation); unit: Total acceptable Words
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 142 | 153 | 180 | 188
Total acceptable Words | -2.0 (9.61) | -0.1 (8.92) | -1.8 (8.12) | -0.8 (8.71)

10. Secondary Outcome: Change From Baseline in Category Fluency Test (CFT)
Description: Study participants are given one minute to provide exemplars of the category 'animals'.
Time Frame: Baseline and 18 months (A-Study); baseline and 12 months (B-Study)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Total Acceptable Words
Arm/Group | A-Study: Azeliragon | A-Study: Placebo | B-Study: Azeliragon | B-Study: Placebo
Number analyzed (Participants) | 142 | 152 | 180 | 188
Total Acceptable Words | -1.7 (4.45) | -1.3 (4.26) | -1.5 (3.80) | 9.7 (146.20)

ADVERSE EVENTS:
Time Frame: Adverse event reporting commenced when the subject received their first dose and ended at the final study visit (21 months).
Groups:
- Azeliragon 5mg: Azeliragon (TTP488) 5mg orally once daily for 18 months
  Parts A and B Combined
- Placebo: Placebo orally once daily for 18 months
  Parts A and B Combined
Arm/Group | Azeliragon 5mg | Placebo
All-Cause Mortality (participants affected / at risk) | 4/441 | 5/434
Serious Adverse Events (participants affected / at risk) | 70/441 | 67/434
Other Adverse Events (participants affected / at risk) | 320/441 | 324/434
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azeliragon 5mg (N=441) | Placebo (N=434)
Syncope (Nervous system disorders) | 4 (4) | 4 (4)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient Ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrage (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 4 (5)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 5 (5)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azeliragon 5mg (N=441) | Placebo (N=434)
Urinary tract infection (Infections and infestations) | 45 (47) | 33 (33)
Nasopharyngitis (Infections and infestations) | 19 (19) | 23 (24)
Upper Respiratory Tract Infection (Infections and infestations) | 20 (23) | 16 (17)
Bronchitis (Infections and infestations) | 9 (9) | 14 (14)
Sinusitis (Infections and infestations) | 9 (9) | 9 (9)
Influenza (Infections and infestations) | 7 (7) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 20 (22)
Nausea (Gastrointestinal disorders) | 14 (14) | 10 (10)
Constipation (Gastrointestinal disorders) | 10 (10) | 8 (8)
Dizziness (Nervous system disorders) | 18 (19) | 15 (15)
Headache (Nervous system disorders) | 15 (16) | 19 (19)
Syncope (Nervous system disorders) | 7 (8) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 48 (59) | 55 (59)
Laceration (Injury, poisoning and procedural complications) | 10 (10) | 11 (13)
Contusion (Injury, poisoning and procedural complications) | 8 (9) | 8 (12)
Depression (Psychiatric disorders) | 21 (21) | 20 (20)
Agitation (Psychiatric disorders) | 14 (16) | 17 (18)
Anxiety (Psychiatric disorders) | 10 (11) | 15 (15)
Insomnia (Psychiatric disorders) | 11 (11) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 14 (14)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (16)
Fatigue (General disorders) | 13 (16) | 14 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 9 (9)
Weight Decreased (Investigations) | 17 (17) | 13 (13)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (5) | 9 (9)
Atrial Fibrillation (Cardiac disorders) | 5 (7) | 7 (8)
Hypertension (Vascular disorders) | 10 (10) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Where PI requires the use of the Study Results for publication, the PI shall seek the Sponsor's written approval which shall not be unreasonably withheld; provided, however, that (i) Sponsor may require removal of any Confidential Information of Sponsor or may delay publication for a reasonable period of time in order to secure protection any IP Rights; and, (ii) as the Study is designed as a multi-center Study, no publication shall be made until after the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT02080364/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT02080364/SAP_001.pdf